CLINICAL TRIAL: NCT00019565
Title: The Use of Positron Emission Tomography (PET) and Magnetic Resonance Imaging (MRI) to Assess the Effects of Anti-neoplastic Therapy on Tumor Associated Vasculature
Brief Title: PET and/or MRI Scans in Assessing Tumor Response in Patients Receiving Antiangiogenesis Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: 980163; 98-C-0163; CDR0000066720; NCT00001709 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

INTERVENTIONS:
Procedure: magnetic resonance imaging
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Diagnostic procedures, such as PET and MRI scans, may help to measure a patient's response to treatment.

PURPOSE: This diagnostic trial is studying how well PET and/or MRI scans work in assessing changes in tumor blood supply in patients receiving antiangiogenesis therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the ability of positron emission tomography (PET) to assess the effect of therapy directed against tumor vasculatures on tumor blood flow and tumor blood volume in patients enrolled on a treatment protocol evaluating a therapeutic modality effecting the tumor associated vasculature.
* Evaluate the ability of PET to assess the effects of this type of therapy regimen on tumor uptake of fluorodeoxyglucose in these patients.
* Evaluate the ability of magnetic resonance imaging (MRI) to assess the effects of therapy directed against the tumor vasculature on tumor blood flow and tumor vascular density in these patients.
* Compare the findings on PET and/or MRI with those obtained from conventional CT in this patient population.

OUTLINE: This is a diagnostic study conducted concurrently with a therapeutic modality study.

Patients have magnetic resonance imaging and/or positron emission tomography (PET) scans performed prior to start of therapy, 6 weeks and 16 weeks following the initiation of therapy, and 6 weeks following the completion of therapy. Each scan requires about 1-3 hours. Patients receive up to 3 different PET scans including tumor blood flow scan with H2015, tumor blood volume scan with 11CO, and glucose uptake scan with fludeoxyglucose F 18.

PROJECTED ACCRUAL: A total of 145 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Eligible for a treatment protocol evaluating a therapeutic modality that may have an effect on tumor associated vasculature
* Measurable or evaluable disease by standard CT or MRI
* At least 1 lesion measuring greater than 2 cm in diameter

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No pacemakers, aneurysm clips, shrapnel injury, or implantable electronic devices
* Weight no greater than 136 kilograms
* No sensitivity to contrast agents that cannot be controlled with premedication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1998-10; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States